CLINICAL TRIAL: NCT04384705
Title: HDL Target of CoViD19 ? Analysis on the Caregivers of the Reunion University Hospital
Acronym: H-Cov-Run
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/CHU/08
Record Dates: First submitted 2020-05-06; First posted 2020-05-12 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: SARS-CoV Infection
MeSH Terms: conditions — Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- caregivers: caregivers
  Interventions: Other: research specific blood sample

INTERVENTIONS:
Other: research specific blood sample — * one blood sample before the epidemic phase
  * one blood sample during epidemic phase
  * one blood sample after epidemic phase

SUMMARY:
Since December 2019, the Severe Acute Respiratory Syndrome-Coronavirus-2 (SARS-CoV-2) pandemic has spread around the world. The people most exposed to this virus remain the healthcare personnel who are on the front line in the fight against this pandemic. Due to the delayed nature of the pandemic in Reunion island and its insular geographical situation, the study of the voluntary medical personnel will allow the investigators to establish a longitudinal follow-up of the anomalies of the lipidic balance in relation to the exposure to the SARS-Cov virus. 2. During bacterial infections, the lipid profiles are profoundly modified with very significant reductions in plasma cholesterol levels, LDL-C but especially HDL-C whose concentrations are particularly low. Lipid profiles are altered during viral infections, for example, the severity of dengue is inversely correlated with total cholesterol and LDL-C but not with HDL-C levels, according to a recent meta-analysis. The hepatitis C virus circulates in serum linked to lipoproteins rich in triglycerides and HDL can facilitate its entry into cells via Scavenger receptor class B type 1 (SRB1). Likewise, it has been shown that apoA1 can bind to the dengue virus and increase its infectivity by promoting its entry into cells, also via SRB1. At the moment, nothing is known about the lipid profiles in subjects with SARS-CoV-2. The investigator hypothesize that a drop in plasma HDL-C levels and a change in their size during infection could justify future therapeutic approaches aimed at supplementing the subjects most at risk of pulmonary complications. In a model of Pseudomonas aeruginosa pneumonia in mice, investigators have shown that the injection of reconstituted HDL allowed to limit the pulmonary inflammation and the deleterious consequences of the infection. The investigator propose to study not only the lipid profiles in subjects who are infected with SARS-CoV-2 but also the polymorphisms of genes involved in the regulation of lipoprotein levels like that of Cholesterol Ester-Transfer Protein (CETP) depending on the developed forms, symptomatic or not.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver in Reunion island University Hospital Center
* Practicing in a care service possibly exposed to the coronavirus
* Signed Consent

Exclusion Criteria:

* Refusal to participate
* Already infected by Covid19

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caregiver in Reunion island University Hospital Center who practice in a care service possibly exposed to the coronavirus
Sampling Method: Non-Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change of lipid profile during exposure to SARS-Cov-2 | at the end of the study, maximum 1 year
  lipid profile

SECONDARY OUTCOMES:
HDL-cholesterol size | at the end of the study, maximum 1 year
  HDL-cholesterol size
circulating plasma cytokine levels | at the end of the study, maximum 1 year
  circulating plasma cytokine levels
ACE2 gene polymorphisms | at the end of the study, maximum 1 year
  ACE2 gene polymorphisms

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire Réunion, Saint-Denis
  - Centre Hospitalier Universitaire de la Réunion, Saint-Pierre

IPD SHARING:
Plan to Share IPD: No